CLINICAL TRIAL: NCT02960100
Title: S.M.A.R.T. (Students Motivating and Acting in Real-Time) eStudy
Brief Title: mHealth Intervention in Increasing HPV Vaccinations in College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mira Katz, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-16109; NCI-2016-01449 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016058 (NIH)
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Healthy Subject
Keywords: Cancer prevention; HPV; Human papillomavirus vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (mHealth HPV vaccine intervention) (Experimental): Participants receive targeted HPV vaccine narrative-style video via the mobile-friendly website. Participants also receive monthly HPV vaccination reminders via email or by text message.
  Interventions: Other: Media Intervention; Other: Survey Administration
- Arm II (standard HPV information and HPV VIS) (Active Comparator): Participants receive standard information with the HPV Vaccine Information Statement via the mobile-friendly website.
  Interventions: Other: Informational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Informational Intervention — Receive standard HPV vaccine information (HPV VIS)
  Arms: Arm II (standard HPV information and HPV VIS)
Other: Media Intervention — Receive targeted HPV vaccine narrative-style video
  Arms: Arm I (mHealth HPV vaccine intervention)
Other: Survey Administration — Ancillary studies

SUMMARY:
This randomized pilot trial studies how well a mobile health (mHealth) intervention works in increasing human papillomavirus (HPV) vaccination among college students at the Ohio State University. mHealth educational intervention may communicate information about HPV vaccination and increase HPV vaccine uptake in college students.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Pilot test an mHealth HPV vaccine intervention for college students to establish feasibility and acceptability.

II. Obtain preliminary efficacy data on whether the mHealth HPV vaccine intervention increases HPV vaccine initiation compared to the control group.

SECONDARY OBJECTIVES:

I. Examine whether the mHealth HPV vaccine intervention affects secondary outcomes compared to the control group.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive targeted HPV vaccine narrative-style video via the mobile-friendly website. Participants also receive monthly HPV vaccination reminders via email or by text message.

ARM II: Participants receive standard information about HPV and then HPV vaccine information statement (VIS) via the mobile-friendly website.

After completion of study, participants are followed up at 3 and 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled as a first year Ohio State University (OSU) student on the Columbus campus
* Being able to read English
* Not having received any doses of the HPV vaccine

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Receipt of the first dose of HPV vaccine in intervention and control group | Up to 7 months
  Will obtain preliminary efficacy data on whether the mHealth HPV vaccine intervention increases HPV vaccine initiation compared to the control group.
Participant satisfaction scores | Up to 7 months
  Acceptability and feasibility will be established by examining participant satisfaction with study materials.

OTHER OUTCOMES:
Receipt of the second and third doses of the HPV vaccine series by intervention and control group | Up to 7 months
  Will examine whether the mHealth HPV vaccine intervention affects the receipt of the second and third doses of the HPV vaccine series compared to the control group.
Changes in potential mediators between intervention or control group and HPV vaccination | Up to 7 months
  Will examine whether the mHealth HPV vaccine intervention affects changes in potential mediators between intervention group and HPV vaccination compared to the control group.
Student feedback based on satisfaction and usability data assessed by surveys | Up to 7 months
Number of times participant logged in to view the narrative or HPV VIS | Up to 7 months
Number of times participants in the intervention group used the link to make an appointment at the health center | Up to 7 months
Total time spent viewing the narrative-style video or HPV VIS | Up to 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Mira Katz, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No